CLINICAL TRIAL: NCT03462771
Title: Effect of Dietary Supplementation With Omega-3 Fatty Acid on the Adaptive Muscular Response to Resistance Training in Sarcopenic Elderly Women
Brief Title: Dietary Supplementation With Omega-3 Fatty Acid in Muscle Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eduardo Ferriolli (Other)
Responsible Party: Sponsor-Investigator, Eduardo Ferriolli, Assistant professor, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 5607/2016
Record Dates: First submitted 2018-02-26; First posted 2018-03-13 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Elderly Women; Sarcopenia
Keywords: elderly; sarcopenia; dietary supplementation; omega-3 fatty acid
MeSH Terms: conditions — Sarcopenia | interventions — Fish Oils; Docosahexaenoic Acids; Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group exercise fish oil (Experimental): Using the Randomizer Research program, 15 elderly women will participate in a resistance exercise protocol and receive omega-3 fatty acid supplements to be ingested 2g in the main meals, totaling 4g daily.
  Interventions: Drug: Fish oil
- Group exercise placebo (Placebo Comparator): Using the Randomizer Research program, 15 elderly women will participate in a resistance exercise protocol and receive sunflower oil to be ingested 2g in the main meals, totaling 4g daily.
  Interventions: Drug: sunflower oil

INTERVENTIONS:
Drug: Fish oil — 4g of fish oil daily for 14 weeks
  Other Names: Omega 3
  Arms: Group exercise fish oil
Drug: sunflower oil — 4g of sunflower oil daily for 14 weeks
  Other Names: Omega 6
  Arms: Group exercise placebo

SUMMARY:
Both aging and other factors associated with it may contribute to the development of sarcopenia, such as lack of physical activity, inadequate food intake, hormonal changes and age-related increases in cytokine levels. What is a growing number of elderly people in Brazil and the world, it is extremely important to conduct research in order to know the mechanisms of action of new strategies to combat sarcopenia. Supplementation with omega-3 fatty acids is a promising intervention in sarcopenic rest. However, there is a practice of studies confirming the effects of omega-3 fatty acid supplementation on neuromuscular function in the elderly.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of omega 3 polyunsaturated fatty acid supplementation on the muscular adaptive response in sarcopenic elderly women submitted to resistance training. A total of 30 sarcopenic elderly women, aged 65 years or older, were divided into two groups of 15 volunteers: (1) Exercise group and placebo (GEP) and (2) Exercise group and fish oil (GEOP). The two groups underwent a resisted exercise program over 12 weeks in three weekly sessions supervised by physicists and physicists at the School of Physical Education and Sports of Ribeirão Preto (EEFERP). All volunteers (both groups) are also instructed to ingest two food supplement capsules at each main meal, and the GEP group will use capsules composed of sunflower oil as a placebo. The GEOP is directed to take two capsules of fish oil at each main meal, totaling 4 capsules per day, that is, four grams of fish oil. To check the quadriceps muscle volume before and after an intervention, as volunteers from both groups are submitted to MRI. An extension power and isokinetic force of extension of the lower limb at a knee and hip extension and are measured by dynamometry (Biodex 4 Pro, Biodex, USA) and a functional solution evaluated by the application of the 6-minute walk test. In addition, will be described the biochemicals for the quantification of the following cytokines: IL1, IL6, IL8, IL10 and TNF-α, such as to allow selection of the presence of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Being sedentary (moderate to vigorous physical activity for at least 3 months)
* BMI <30.00 kg / m2;

Exclusion Criteria:

* Any type of absolute and / or relative contraindication to moderate or intense physical activity.
* Any physical limitation that makes it impossible to practice physical activities and / or that impairs the performance of the tests.
* Also not included are those volunteers who do not go through pre-Physical Activity evaluation. (Par Q Questionnaire)
* miss more than 3 workouts consecutive

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-21 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline muscle volume after 14 weeks | before and after 14 weeks
  Calculated by Nuclear Magnetic Resonance
Change from Baseline muscle strength of knee extensors after 14 weeks | before and after 14 weeks
  Measure of muscle strength of the lower limbs (knee extension) with a isokinetic dynamometer (Biodex 4 Pro)

SECONDARY OUTCOMES:
Assessment of serum levels of inflammatory cytokines | before and after 14 weeks
  Evaluated by blood samples
Assessment of physical performance | before and after 14 weeks
  The physical performance will be evaluated by the Short Physical Performance Battery test.
Assessment of handgrip strength | before and after 14 weeks
  Measure of handgrip strength with a manual dynamometer (Saehan)
Physical Activity behaviour | before and after 14 weeks
  use of a tri-axial accelerometer to measure profile of spontaneous physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ferriolli, PhD, Principal Investigator — University of Sao Paulo; Carolyn Greig, Study Chair — University of Birmingham
Locations (1):
- Clinics Hospital of the Ribeirao Preto Medical School Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Da Boit M, Sibson R, Sivasubramaniam S, Meakin JR, Greig CA, Aspden RM, Thies F, Jeromson S, Hamilton DL, Speakman JR, Hambly C, Mangoni AA, Preston T, Gray SR. Sex differences in the effect of fish-oil supplementation on the adaptive response to resistance exercise training in older people: a randomized controlled trial. Am J Clin Nutr. 2017 Jan;105(1):151-158. doi: 10.3945/ajcn.116.140780. Epub 2016 Nov 16. PMID 27852617